CLINICAL TRIAL: NCT01729988
Title: Carotid Body Removal for the Treatment of Resistant Hypertension: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noblewell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBR-GDAPL-CIBIEM
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carotid body excision (Experimental): Patients undergoing the carotid body excision to test the hypothesis that carotid body excision is sufficient to attain target blood pressure.
  Interventions: Procedure: Carotid body excision

INTERVENTIONS:
Procedure: Carotid body excision — This surgery does not involve any study drug or investigational device.
  The carotid body will be removed by the so called 'lateral approach' or a combined 'lateral and medial approach'. In all cases the target area was defined as the tissue in between the ECA and ICA, up to 5-6mm above the bifurcation point of the common carotid artery into the ECA and ICA. In a lateral approach the carotid bifurcation is not turned. A combined approach includes usually dissection of the superior thyroid vessel and turning of the carotid bifurcation.

SUMMARY:
This is a pilot study to assess the effectiveness, safety and feasibility of carotid body removal in patients with high blood pressure (hypertension) resistant to medical treatment. Patients with high blood pressure are at significant risk of medical complications including stroke and heart disease. The principle research question is whether removal of the carotid body will lead to an improvement in the blood pressure of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Resistant HTN criteria with either confirmed sleep disordered breathing. Definition of HTN:Office SBP ≥ 160 mmHg and daytime mean ABPM ≥ 140 mm Hg
* Definition of sleep disordered breathing: SDB defined as mild to moderate obstructive, central or mixed sleep apnea defined as 5 < AHI < 30 with O2 desaturation not exceeding 80% during the night.

Exclusion Criteria:

* Calculated GFR < 30
* Carotid body located outside the defined carotid septum
* Obstructive carotid atherosclerotic disease
* Oxygen desaturation at rest below 92%
* Known structural lung disease (medical interview)
* Requirement for oxygen therapy to maintain oxygen saturation
* Patients wish to participate in mountain climbing, skin diving or free diving
* Pregnancy or anticipation of pregnancy
* Palliative care/chemotherapy
* Acute coronary syndrome or unstable angina < 6 months prior to procedure
* Use of exogenous insulin AND history of hypoglycemic unawareness
* Stroke or transient ischaemic attack (TIA), or myocardial infarction < 6 months prior to procedure
* Expected life expectancy less that 24months due to other disease
* Intravenous drug use
* Excessive use of alcohol or sedatives (Alcohol intake >28 units/week)
* Obesity (BMI > 40)
* Upper airway or facial abnormalities
* Large neck circumference (>43.2 cm men; >40.6 cm women)
* Febrile illness within two weeks of participation
* Unable to attend for follow up appointments at 1, 3 and 6 months post operatively.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change of Blood Pressure | 3 months
  Change from Baseline Blood Pressure at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Sobotka, M.D., Study Director — Cibiem, Inc.
Locations (1):
- Department of Hypertension and Diabetology, Medical University of Gdansk, Gdansk, Poland